CLINICAL TRIAL: NCT03113227
Title: Diagnostic Accuracy of Posterior Cervical Angle and Cervical Length in Prediction of Successful Induction of Labor
Brief Title: Value of Measuring Cervical Angle and Length by Ultrasound in Prediction of Successful Induction of Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Omran, Principal investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 5355
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Induced; Birth
Keywords: induction of labor; Bishop score; posterior cervical angle; cervical length
MeSH Terms: interventions — Gynecological Examination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Successful Induction of labor group (Active Comparator): Both transvaginal ultrasound and vaginal examination will be done for that group
  Interventions: Diagnostic Test: Transvaginal ultrasound; Diagnostic Test: Vaginal examination
- Failed induction of labor group (Active Comparator): Both transvaginal ultrasound and vaginal examination will be done for that group
  Interventions: Diagnostic Test: Transvaginal ultrasound; Diagnostic Test: Vaginal examination

INTERVENTIONS:
Diagnostic Test: Transvaginal ultrasound — Transvaginal ultrasound will be made for assessment of posterior cervical angle and cervical length
Diagnostic Test: Vaginal examination — Vaginal examination will be done for assessment of Bishop score

SUMMARY:
Seventy ladies indicated for induction of delivery will be recruited. Two ways of assessment of their cervices will be done before actual induction of labor. First, ultrasound will be done to assess the angle and the length of the cervix. Then vaginal examination will be done to assess the characteristics of cervix. Analysis will be done to identify the best predictor of successful induction of labour.

DETAILED DESCRIPTION:
Seventy patients indicated for induction of labor will be recruited. Two ways of assessment of their cervices will be done before actual induction of labor. First, transvaginal ultrasound will be done to assess the posterior angle and the length of the cervix. Then vaginal examination will be done to measure the Bishop score. Analysis will be done to identify the best predictor of successful induction of labour.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestational age between 35 and 42
* Presence of an indication for induction of labour as post-term pregnancy or rupture of membranes
* The fetus is living
* Cephalic presentation

Exclusion Criteria:

* Estimated fetal weight more than 4 kilograms
* Malpresentation
* Oligohydramnios
* Polyhydramnios
* Non-reassuring non-stress test before induction of labor
* Cephalo-pelvic disproportion
* Previous operation on the cervix as cautery or cerclage
* Previous cesarean section
* Any contraindication to vaginal delivery including placenta previa
* Anomalous fetus
* Morbid obesity

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2017-07-09 (Actual); Study Completion 2017-07-09 (Actual)

PRIMARY OUTCOMES:
Value of posterior cervical angle | At around 10 minutes from admission to hospital
  Value of posterior cervical angle will be measured by an investigator

SECONDARY OUTCOMES:
Length of the cervix | At around 10 minutes from admission to hospital
  Length of the cervix will be measured by an investigator
Bishop score | At around 30 minutes from admission to hospital
  Bishop score will be measured by an investigator

CONTACTS AND LOCATIONS:
Overall Officials: Eman Omran, M.D., Principal Investigator — Cairo University
Locations (1):
- Department of Obstetrics and Gynecology, Kasr Al-Ainy hospital, Cairo, Greater Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Al-Adwy AM, Sobh SM, Belal DS, Omran EF, Hassan A, Saad AH, Afifi MM, Nada AM. Diagnostic accuracy of posterior cervical angle and cervical length in the prediction of successful induction of labor. Int J Gynaecol Obstet. 2018 Apr;141(1):102-107. doi: 10.1002/ijgo.12425. Epub 2018 Jan 18. PMID 29224196